CLINICAL TRIAL: NCT06724809
Title: An Open-label, Single-arm, Multi-Center, Interventional Study to Evaluate the Efficacy, Safety, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Eculizumab in Chinese Adult Participants With Anti-Aquaporin-4 Antibody Positive Neuromyelitis Optica Spectrum Disorders (NMOSD)
Brief Title: Efficacy, Safety, PK, PD, and ADA of Eculizumab in Chinese Adults With NMOSD
Acronym: ECU-NMO-304
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D7412C00002
Record Dates: First submitted 2024-11-19; First posted 2024-12-09 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: NMOSD; Neuromyelitis Optica Spectrum Disorders
Keywords: NMOSD; Neuromyelitis Optica Spectrum Disorders; eculizumab; anti-AQP4
MeSH Terms: conditions — Neuromyelitis Optica | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- eculizumab (Experimental): All participants will receive open-label eculizumab by intravenous infusion during the Treatment Period, starting on Day 1 for a total of up to 52 weeks.
  Interventions: Drug: eculizumab

INTERVENTIONS:
Drug: eculizumab — Participants will receive eculizumab by intravenous (IV) infusion for 52 weeks.

SUMMARY:
The primary objective of this study is to evaluate the efficacy, safety, pharmacokinetics, pharmacodynamics, and immunogenicity of Eculizumab in Chinese Adults with Neuromyelitis Optica Spectrum Disorders (NMOSD).

ELIGIBILITY:
Inclusion Criteria:

* Participants with diagnosis of NMOSD as defined by the 2015 international consensus diagnostic criteria
* Anti-AQP4 antibody positive
* At least 1 attack or relapse in the last 12 months prior to the Screening Period
* EDSS score ≤ 7
* If a participant enters the study receiving IST(s) for relapse prevention, the participant must be on a stable maintenance dose of IST(s) as follows, prior to screening and must remain on that dose for the duration of the study, unless the participant experiences a relapse
* Female participants of childbearing potential must have a negative pregnancy test (serum HCG at screening
* Male participants are eligible to participate if they agree to the following during the study intervention Treatment Period and for at least 5 months after the last dose of study intervention:

  * Refrain from donating fresh unwashed semen. PLUS, either,
  * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent. OR
  * Must agree to use barrier as detailed below:

    * Agree to use a male condom when having sexual intercourse with a WOCBP who is not currently pregnant.

Exclusion Criteria:

* Pregnant, breastfeeding, or intending to conceive during the course of the study
* Prior history of N meningitidis infection or unresolved meningococcal disease
* Any systemic bacterial or other infection which is clinically significant in the opinion of the Investigator and has not been treated with appropriate antibiotics
* Presence of fever ≥ 38 C within 7 days prior to study intervention administration on Day 1
* Hypersensitivity to murine proteins or to one of the excipients of study intervention
* Use of rituximab, inebilizumab, or other B cell-depleting therapy within 6 months prior to Day 1 and during the study
* Use of mitoxantrone or satralizumab within 3 months prior to screening and during the study
* Use of IVIg within 3 weeks prior to screening
* If a participant enters the study receiving oral corticosteroid(s) with or without other ISTs, the daily corticosteroid dose must be no more than prednisone 20 mg/day (or equivalent) prior to screening and the participant must remain on that dose for the duration of the study or until the participant experiences a relapse (specific medications listed in Section 6.9.1 may be allowed)
* Has previously received treatment with C5 inhibitors
* Participation in any other investigational drug study or exposure to an investigational drug or device within 5 half-lives of treatment (if known) or 30 days, which is longer, before the first dose administration

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2025-01-16 (Actual); Primary Completion 2026-12-07 (Estimated); Study Completion 2026-12-07 (Estimated)

PRIMARY OUTCOMES:
The efficacy of eculizumab in anti-AQP4 antibody positive participants with NMOSD measured by Adjudicated On-trial annualized relapse rate (ARR). | Baseline through Week 52
  The mean (95% Confidence Interval) of patient-level Adjudicated On-trial annualized relapse rate (ARR)
The efficacy of eculizumab in anti-AQP4 antibody positive participants with NMOSD measured by Adjudicated On-trial annualized relapse rate (ARR). | Baseline through Week 52
  Intercurrent Event (ICE):
  * ICE1: Premature discontinuation of study intervention
  * ICE2: Initiation of disallowed therapy or medicine

SECONDARY OUTCOMES:
The efficacy of eculizumab by assessing change from baseline to end of study in Expanded Disability Status Scale (EDSS) Score | Baseline through Week 52
  Intercurrent Event (ICE):
  * ICE1: Premature discontinuation of study intervention
  * ICE2: Initiation of disallowed therapy or medicine
    * Summary measure: The mean (95% Confidence Interval) change from baseline to end of study in EDSS score
The efficacy of eculizumab by assessing change from baseline to end of study in Ambulatory Function as Measured by Hauser Ambulation Index (HAI) | Baseline through Week 52
  Intercurrent Event (ICE):
  * ICE1: Premature discontinuation of study intervention
  * ICE2: Initiation of disallowed therapy or medicine
    * Summary measure: The mean (95% Confidence Interval) change from baseline to end of study in ambulatory function as measured by Hauser ambulation index (HAI)
The efficacy of eculizumab by assessing change from baseline to end of study in European Quality of Life 5-Dimension Questionnaire (EQ-5D) Index Score | Baseline through Week 52
  Intercurrent Event (ICE):
  * ICE1: Premature discontinuation of study intervention
  * ICE2: Initiation of disallowed therapy or medicine
    * Summary measure: The mean (95% Confidence Interval) change from baseline to end of study in EQ-5D index score
Change From Baseline to end of study in EQ-5D Visual Analogue Scale (VAS) Score | Baseline through Week 52
  Intercurrent Event (ICE):
  * ICE1: Premature discontinuation of study intervention
  * ICE2: Initiation of disallowed therapy or medicine
    * Summary measure: The mean (95% Confidence Interval) change from baseline to end of study in EQ-5D VAS
Serum Eculizumab Concentrations Over Time | Baseline through Week 52
  Intercurrent Event (ICE):
  * ICE1: Premature discontinuation of study intervention
  * ICE2: Initiation of disallowed therapy or medicine
    * Summary measure: Mean serum eculizumab concentrations at all scheduled visits
Serum Free Complement Component 5 (C5) Concentrations Over Time | Baseline through Week 52
  Intercurrent Event (ICE):
  * ICE1: Premature discontinuation of study intervention
  * ICE2: Initiation of disallowed therapy or medicine
    * Summary measure: Mean changes in serum free C5 concentrations at all scheduled visits
Number of Treatment-emergent Antidrug Antibody (ADA) Positive Participants | Baseline through Week 52
  Intercurrent Event (ICE):
  * ICE1: Premature discontinuation of study intervention
  * ICE2: Initiation of disallowed therapy or medicine
    * Summary measure: Proportion of treatment-emergent ADA positive participants
To characterize the overall safety of eculizumab in the treatment of NMOSD | Baseline through Week 52
  Number of participants with TEAEs, SAEs, and TEAEs leading to study intervention discontinuation, with abnormal vital signs, abnormal ECG readings, and abnormal laboratory tests results

CONTACTS AND LOCATIONS:
Overall Officials: Xiangjun Chen, M.D, Principal Investigator — Huashan Hospital
Locations (7):
- China (7):
  - Research Site, Beijing
  - Research Site, Dongguan
  - Research Site, Jinan
  - Research Site, Shanghai
  - Research Site, Taiyuan
  - Research Site, Wenzhou
  - Research Site, Wuhan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home